CLINICAL TRIAL: NCT01765478
Title: A Phase1 Study, to Determine the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of Single and Multiple Doses of Orally Administered HM71224 in Healthy, Adult Male Volunteers
Brief Title: Safety,PK/PD, Food Effect Study of Orally Administered HM71224 in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-HM71224-101
Record Dates: First submitted 2013-01-07; First posted 2013-01-10 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2012-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (11):
- Treatment A Period 2 (Experimental): 40mg HM71224 single dose
  Interventions: Drug: HM71224 single ascending dose
- Treatment B Period1 (Experimental): 20mg HM71224 single dose
  Interventions: Drug: HM71224 single ascending dose
- Treatment A Period1 (Experimental): 10mg HM71224 single dose
  Interventions: Drug: HM71224 single ascending dose
- Treatment B Period2 (Experimental): 80mg HM71224 single dose
  Interventions: Drug: HM71224 single ascending dose
- TreatmentA Period3 (Experimental): 160mg HM71224 single dose
  Interventions: Drug: HM71224 single ascending dose
- TreatmentB Period3 (Experimental): 200mg HM71224 single dose
  Interventions: Drug: HM71224 single ascending dose
- Food effect period1 (Experimental): active 4subjects + placebo 4subjects
  Interventions: Drug: HM71224 food effect
- Food effect period2 (Experimental): active 4subjects + placebo 4subjects
  Interventions: Drug: HM71224 food effect
- TreatmentC (Experimental): HM71224 Xmg multiple dose for 14days
  Interventions: Drug: HM71224 Multiple ascending dose
- TreatmentD (Experimental): HM71224 Ymg 14days multiple dose
  Interventions: Drug: HM71224 Multiple ascending dose
- TreatmentE (Experimental): HM71224 Zmg 14days multiple dose
  Interventions: Drug: HM71224 Multiple ascending dose

INTERVENTIONS:
Drug: HM71224 single ascending dose
  Arms: Treatment A Period 2; Treatment A Period1; Treatment B Period1; Treatment B Period2; TreatmentA Period3; TreatmentB Period3
Drug: HM71224 food effect
  Arms: Food effect period1; Food effect period2
Drug: HM71224 Multiple ascending dose
  Arms: TreatmentC; TreatmentD; TreatmentE

SUMMARY:
HM71224 is a potent small molecule inhibitor of Bruton's tyrosine kinase (BTK). BTK is a member of the Tec family of non-receptor protein tyrosine kinases. BTK is mostly expressed in hematopoietic cells such as B cells, mast cells and macrophages. BTK plays key roles in multiple cell signaling pathways including B-Cell Receptor (BCR) and Fc receptor (FcR) signaling cascades and is an essential mediator not only in B-cell dependent but also in myeloid cell dependent inflammatory arthritis. HM71224 has been selected as a novel therapeutic agent for the treatment of autoimmune diseases such as rheumatoid arthritis (RA).

In view of the above, further development of HM71224 for the treatment of RA is warranted. In this first-in-man (FIM) study, a single and multiple dose escalation design will be employed, in which the primary objective is to evaluate the safety and tolerability of the compound. The biomarkers included as pharmacodynamic (PD) variables are chosen as they are indicators for any effects of HM71224 on the expected mode of action (pBTK, pPLCγ, and pERK).

DETAILED DESCRIPTION:
Primary objective

* To evaluate the safety and tolerability, and if possible maximum tolerated dose (MTD) of HM71224 after single and multiple ascending dose administration in healthy subjects.

Secondary objective

* To determine the PK of HM71224 and selected metabolites (M1 and M2) following single and multiple oral dose administration of HM71224.
* To assess the PD effects of HM71224 on the biomarkers pBTK, pPLCγ, and pERK.
* To assess whether the PK of HM71224 is affected by food.

ELIGIBILITY:
Inclusion Criteria:

1. Gender : male
2. Age : 18-65 years, inclusive
3. BMI : 18.5 - 30.0 kg/m2
4. Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, energy drinks), and grapefruit (juice) from 48 h prior to entry in the clinical research center until discharge
5. Medical history without major pathology
6. Normal resting supine blood pressures and pulse rate, showing no clinically relevant deviations as judged by the MI
7. Computerized (12-lead) electrocardiogram (ECG) recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the MI
8. Willingness to use adequate contraception from the time of dosing until 90 days after the follow-up visit
9. All values for hematology and for clinical chemistry tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the MI
10. Willingness to sign the written Informed Consent Form (ICF)

Exclusion Criteria:

1. Previous participation in the current study
2. Evidence of clinically relevant pathology
3. Mental handicap
4. History of relevant drug and/or food allergies
5. Regular/routine treatment with non-topical medications within 30 days prior to entry into the clinical research center
6. Use of tobacco products within 60 days prior to drug administration
7. History of alcohol abuse or drug addiction (including soft drugs like cannabis products)
8. Use of concomitant medication, except for acetaminophen (paracetamol), which is allowed up to 3 days before entry into the clinical research center. Multivitamins and vitamin C are allowed up to 7 days before entry into the clinical research center. All other medication (including over the counter medication, health supplements, and herbal remedies such as St. John's Wort extract) must have been stopped at least 14 days prior to entry into the clinical research center. The use of a limited amount of acetaminophen during the study is permitted.
9. Participation in a drug study within 60 days prior to drug administration. Participation in more than 3 other drug studies in the 10 months preceding the start of this study (this is the first administration of study drug).
10. Donation of more than 50 mL of blood within 60 days prior to drug administration. Donation of more than 1.5 liters of blood in the 10 months preceding the start of this study (this is the first administration of study drug).
11. Positive drug screen (opiates, methadone, cocaine, amphetamines, cannabinoids, barbiturates, benzodiazepines, and alcohol)
12. Intake of more than 24 units of alcohol per week (one unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
13. Positive screen on Hepatitis B Surface Antigen (HBsAg), anti-Hepatitis C Virus (HCV) or anti-Human Immunodeficiency Virus (HIV) 1/2
14. Illness within 5 days prior to the first drug administration
15. Non-willingness to consume the FDA breakfast (Part B only)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
To investigate safety and tolerability | 3days
  Number of participants with AE occurrence, clinically significant clinical lab,vital sign, and/or ECG change.

SECONDARY OUTCOMES:
To determine plasma PK parameters | 3days
  Cmax, C trough, tmax, kel, t1/2, AUC, CL/F, Vz, Rac, Ae, CLr, Fe% of HM71224 and selected metabolites M1, M2 following single and multiple oral dose administration of HM71224
To determine urine PK parameters | 3days
  Cmax, C trough, tmax, kel, t1/2, AUC, %AUC, CL/F, Vz, Rac, Ae, CLr, Fe% of of HM71224 and selected metabolites M1, M2 following single and multiple oral dose administration of HM71224

CONTACTS AND LOCATIONS:
Overall Officials: Salah Hadi, MD MSc, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA Clinical research center, Zuidlaren, Netherlands

REFERENCES:
- [Derived] Byun JY, Koh YT, Jang SY, Witcher JW, Chan JR, Pustilnik A, Daniels MJ, Kim YH, Suh KH, Linnik MD, Lee YM. Target modulation and pharmacokinetics/pharmacodynamics translation of the BTK inhibitor poseltinib for model-informed phase II dose selection. Sci Rep. 2021 Sep 21;11(1):18671. doi: 10.1038/s41598-021-98255-7. PMID 34548595